CLINICAL TRIAL: NCT04166006
Title: A Phase II Study on Adjuvant Vaccination with Dendritic Cells Loaded with Autologous Tumor Homogenate in Resected Stage IV Rare Cancers: Head&Neck (H&N), Neuroendocrine Tumors (NET) and Soft Tissue Sarcoma (STS).
Brief Title: A Phase II Study on Adjuvant Vaccination with Dendritic Cells Loaded with Autologous Tumor Homogenate in Resected Stage IV Rare Cancers.
Acronym: RaC-Ad
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST100.42
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Head Neck Tumors; Neuroendocrine Tumors; Soft Tissue Sarcoma; Rare Cancer; Vaccination
Keywords: Head Neck Tumors; Neuroendocrine Tumors; Soft Tissue Sarcoma; rare cancer; vaccination; autologous dendritic cells; adjuvant; Interleukin-2
MeSH Terms: conditions — Head and Neck Neoplasms; Neuroendocrine Tumors; Sarcoma | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): 7-14×106 autologous dendritic cells loaded with autologous tumour homogenate given by intradermal injection (day 1), followed by Interleukin (IL) - 2 (IL-2), at a dose of 3 Million Units (MU), given by subcutaneous injection daily for five days (days 3-7). This constitutes a treatment cycle.
  Treatment cycles are repeated every 28 days up to a maximum of six cycles.
  Interventions: Biological: Autologous DC vaccine; Drug: Interleukin-2

INTERVENTIONS:
Biological: Autologous DC vaccine — 7-14×106 autologous dendritic cells loaded with autologous tumour homogenate given by intradermal injection (day 1)
Drug: Interleukin-2 — Autologous DC vaccine is followed by IL-2, at a dose of 3 MU, given by subcutaneous injection daily for five days (days 3-7).

SUMMARY:
Single-arm, monocentric trial to assess safety and immunological efficacy of adjuvant vaccination with autologous dendritic cells loaded with autologous tumour homogenate after curative resection for stage IV rare cancers (In Head/Neck tumors (H&N), NEuroendocrine Tumors (NET) and Soft Tissue Sarcomas (STS).

DETAILED DESCRIPTION:
This is a single-arm, multi-cohort phase II study, to evaluate the immunological effectiveness and safety of adjuvant Dendritic Cell (DC) vaccination. The evaluation of immunological efficacy will be expressed as the number of patients who show enhancement of the proportion of circulating immune effectors specific for a selected panel of associated antigens for each disease (HNSCC, NET and STS). To avoid unacceptable toxicity, a formal safety analysis will be conducted after six patients have been observed (two for each disease) for at least 30 days after the third treatment cycle. If two or more patients have experienced grade 3 or higher adverse events, enrollment will be definitively stopped; differently, other 15 patients for each disease will be enrolled and evaluation of primary objectives will be done for each cohort separately (H&N, STS and NET).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed stage IV Head&Neck Squamous Cell Carcinoma (HNSCC), NeuroEndocrine Tumors (NET) or Soft Tissue Sarcoma (STS) surgically treated with radical intent.
2. The autologous surgical specimen must have been collected and sent to the Somatic Cell Therapy Lab and must fulfil all the acceptance criteria prescribed by the Good Manufactory Practice (GMP) procedures.
3. The patient must be disease-free, as assessed by CT scan or MRI of the chest, abdomen, pelvis performed within 60 days before enrolment. If the resected lesions occurred in other sites, these must be also included in the baseline CT scan and in all the subsequent evaluations.
4. Patients disease-free candidates for only observation as per clinical practice (no standard treatment is available after surgery)
5. The patient must have recovered from all the adverse events related to previous surgery.
6. Age ≥18 years.
7. Performance status Eastern Cooperative Oncology Group (ECOG) 0 or 1.
8. Patient must have acceptable organ function, defined as:

   1. Haemoglobin >10 g/dl
   2. White blood cells ≥3000/μl.
   3. Absolute neutrophil count ≥1500/μl.
   4. Platelets≥75000/μl.
   5. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 times the upper institutional reference level.
   6. Total bilirubin <1.5 times the upper institutional reference level.
   7. Serum creatinine <1.5 times the upper institutional reference level.
9. Patients aged 70 years or older must have left ventricular ejection fraction not lower than 55% as assessed by echocardiography.
10. Female patients of childbearing potential and all male patients must accept and be compliant with an highly effective contraceptive method (i.e. with a failure rate of <1% per year: double barrier method, one barrier method plus spermicidal, intrauterine device, or oral contraception) from informed consent signature and up to three months after end of study. For this purpose are considered of childbearing potential all female subjects after puberty unless they are post-menopausal for at least two years or are surgically sterile. Complete abstinence from sexual intercourses is acceptable if patients' lifestyle guarantees his/her strict compliance with this prescription in the judgement of the Investigator.
11. The patient is willing and able to give written informed consent for the study.

Exclusion Criteria:

1. Patients with residual disease after surgery. Marginal resection of any lesion in the absence of clinically evident residual disease is acceptable.
2. Patient who completed surgery more than 90 days before study enrolment.
3. History of other neoplastic diseases in the previous 5 years, except basal cell carcinoma of the skin and in situ carcinoma of the cervix uteri treated with curative surgery.
4. History of congenital or acquired immunodeficiency, including history of organ transplantation.
5. Any positivity for the serologic markers of hepatitis B virus (HBV) (including at least anti- Hepatitis B surface antibodies (HBs) and hepatitis B core (HBc) antibodies, hepatitis C virus (HCV), HIV or Treponema pallidum. The serologic tests must have been performed within 30 days before any GMP-regulated activity (i.e. surgical resection and leukapheresis). The sole positivity for antibodies against the HBV surface antigen (i.e.

   with all other HBV markers negative) is indicative of previous HBV vaccination and therefore is acceptable.
6. Female patients who are pregnant or nursing.
7. Participation in another clinical trial with any investigational agent within 30 days prior to study screening.
8. Any active inflammatory or autoimmune disease requiring systemic steroids or other immunomodulatory agents as detailed in section 6.4, or potentially requiring such treatments during the study treatment in the judgement of the Investigator.
9. Any clinical condition that, in the opinion of the Investigator or the Transfusion Medicine specialist, is a contraindication to leukapheresis. In addition, all patients aged 70 or older must be evaluated by a cardiology specialist before the procedure to exclude any clinically relevant cardiac condition and any grade 3-4 cardiac arrhythmia, even if asymptomatic.
10. Any uncontrolled serious intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations potentially impacting patient safety and compliance in the opinion of the Investigator.
11. Refusal of giving written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | from the day of the leukapheresis up to 30 days after the last dose
  Incidence, type and severity of adverse events occurred during treatment will be reported and graded according to NCI CTCAE 5.0 criteria
Immunological efficacy | at 4 months, after at least 3 vaccinations
  immunological efficacy will be assessed as a proportion of tumor-specific circulating immune effectors determined by IFNgamma ELISPOT

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 7 years
  OS is the time from registration to the time of death from any cause. Subjects who are alive at the time of the final analysis or who have become lost to follow-up will be censored at their last known alive date.
Relapse Free Survival (RFS) | Up to 7 years
  RFS is the time from registration to the first date of documented progression (or death for any causes). Subject without progression will be censored at their last tumor assessment date.
Predictive role of Delayed-Type Hypersensitivity (DTH) skin test | Up to 7 years
  Evaluation of the predictive role of a positive DTH test after at least three vaccine administrations

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ridolfi, MD, Study Chair — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)
Locations (1):
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC, Italy